CLINICAL TRIAL: NCT00590967
Title: A Phase II Study of Extended Field IMRT External Beam Irradiation and Intracavitary Brachytherapy With Concurrent Weekly Cisplatin in Patients With Stage I-IVA Cervical Cancer Who Have FDG PET Positive Pelvic or Para-Aortic Lymph Nodes
Brief Title: A Phase II Study of Extended Field IMRT External Beam Irradiation and Intracavitary Brachytherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-0300 / 201105362
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-06

CONDITIONS: Cervical Cancer
Keywords: para-aortic lymph nodes
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental): Pelvic Lymph Nodes Only Positive on FDG PET.
  IMRT External Beam radiation to the para-aortic region (45 Gy)
  Pelvis intracavitary brachytherapy (6 HDR treatments)
  Weekly cisplatin 40 mg/m^2
  Interventions: Radiation: IMRT extended field external beam radiation therapy; Radiation: Brachytherapy; Drug: Cisplatin
- Treatment Group 2 (Experimental): Para-Aortic Lymph Nodes Positive on FDG PET
  IMRT (50.4 Gy to para-aortic lymph node bed with a 10.8 Gy boost to nodes)
  IMRT external beam pelvic radiation therapy as appropriate for stage
  Intracavitary brachytherapy (6 HDR treatments)
  Weekly cisplatin (40 mg/m^2)
  Interventions: Radiation: IMRT extended field external beam radiation therapy; Radiation: Brachytherapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: IMRT extended field external beam radiation therapy
Radiation: Brachytherapy
Drug: Cisplatin

SUMMARY:
Recent studies have shown that the chance of survival among women with advanced cervical cancer is increased when they receive concurrent chemotherapy and radiation to the pelvis. However, patients who have advanced disease show loco-regional failure as well as a high incidence of distant metastasis. Positron emission tomography (PET) scanning has high sensitivity and specificity in the detection of pelvic and para-aortic lymph node metastases. While the detection of para-aortic metastases by PET significantly impacts prognosis, PET has been known to show positive lymph node metastasis in the pelvis only while not detecting micrometastatic disease in the para-aortic lymph nodes (despite the fact that they are histologically known).

In addition, patients with positive para-aortic lymph nodes on PET, greater amounts (more than 45 Gy) of radiation must be used to improve the probability of controlling the cancer. However, doses greater than this have been limited because of the dose and volume limits to the small bowel. But, Intensity Modulated Radiation Therapy (IMRT) is a new way of calculating and delivering radiation therapy. Compared to external beam radiation, IMRT has the improved ability to deliver large doses of radiation to specific targets while minimizing the exposure to surrounding normal tissue.

With IMRT, however, the effective dose/volume can be increased more safely and lower the toxicity of surrounding tissue, thus making prophylactic dosing to para-aortic lymph nodes not detected by PET safer and more effective.

DETAILED DESCRIPTION:
Prior to entrance on the study, patients will undergo a history and physical and evaluation of Karnofsky Performance Status. They will have a biopsy of their tumor and will undergo a fluorodeoxyglucose (FDG) PET scan and must include evaluation of para-aortic lymph nodes. Blood work will be done (complete blood count (CBC), differential, platelets, blood urea nitrogen(BUN), serum creatinine, bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase. Also, pre-treatment, patients will receive a chest x-ray and an intravenous push (IVP) (unless a computed tomography (CT) with contrast has been performed). Additionally, patient may undergo a CT, magnetic resonance (MRI) and/or lymphangiogram.

Patients will then be registered to a treatment arm, depending on the outcome of their PET scan. Patients with positive pelvic lymph nodes but no positive para-aortic lymph nodes by PET will be assigned to Treatment Arm 1. Patients with positive pelvic lymph nodes and positive para-aortic lymph nodes by PET will be assigned to treatment arm 2.

Treatment Group 1. Either a conventional or CT simulation may be performed. Patients will be treated with IMRT extended field external beam radiation therapy (to cover pelvis and para-aortic lymph nodes) and intracavitary radiation (6 high dose radiation (HDR) treatments) concurrently with cisplatin (40 mg/m^2/week)

Treatment Group 2. A CT simulation must be performed. Patients will be treated with extended field external beam radiation therapy to the pelvis and with IMRT to cover the para-aortic lymph nodes to 60 Gy, 50.4 Gy to the para-aortic lymph node bed in conjunction with external beam pelvic radiation therapy as appropriate for disease stage and intracavitary radiation (6 HDR treatments) concurrently with cisplatin (40 mg/m^2/week).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have carcinoma of the uterine cervix.
* Patients with squamous cell, adenocarcinoma, and adenosquamous carcinoma are eligible.
* International Federation of Gynecology and Obstetrics (FIGO) Stage I to IVA
* Patients must have no evidence of metastatic disease outside of the pelvis (except to the para-aortic nodes), by PET.
* Patients must have a Karnofsky Performance Status of >= 60 and no medical contraindications to the administration of chemotherapy.
* Age >= 18.
* Adequate bone marrow function: white blood cells (WBC) >= 4000/mm3, platelets >= 100,000 mm3.
* Adequate renal function: BUN <= 25 mg/dl, creatinine <= 1.2 mg/dl (urinary diversion is permitted to improve renal function).
* Patients must have bilirubin <= 1.5 mg/dl.
* Signed study-specific informed consent.

Exclusion Criteria:

* No positive lymph nodes by FDG PET
* Positive supraclavicular lymph nodes by FDG PET Scan or evidence of more distant disease.
* FIGO Stage IVB+ Cervical Cancer
* No prior (within 5 years) or simultaneous malignancies (other than cutaneous basal cell carcinoma).
* Karnofsky Performance Status <60.
* Patients with significant medical illness preventing the use of full dose chemotherapy are excluded.
* Patients with the following histologies are excluded: small cell, carcinoid, glassy cell, clear cell and adenoid cystic.
* Life expectancy < 6 months.
* Patients with poorly controlled diabetes mellitus (fasting blood glucose level > 200 mg/dL) are not eligible.
* No prior surgery for treatment of disease other than exploratory laparotomy or biopsy.
* No previous systemic chemotherapy.
* No pelvic radiation therapy is permitted other than transvaginal irradiation to control bleeding.
* Pregnant women are ineligible and those of child-bearing potential should practice contraception.
* Patients with abnormal liver function tests

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Grigsby, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to patient accrual on 05/01/2003 and closed to patient accrual on 04/24/2008.
Groups:
- Treatment Group 1 (IMRT, Brachytherapy, Cisplatin): Pelvic Lymph Nodes Only Positive on fluorodeoxyglucose (FDG) positron emission tomography (PET).
  Intensity-modulated radiation therapy (IMRT) External Beam radiation to the para-aortic region (45 Gy)
  Pelvis intracavitary brachytherapy (6 high dose radiation (HDR) treatments)
  Weekly cisplatin 40 mg/m^2
- Treatment Group 2 (IMRT, Brachytherapy, Cisplatin): Para-Aortic Lymph Nodes Positive on FDG PET
  IMRT (50.4 Gy to para-aortic lymph node bed with a 10.8 Gy boost to nodes)
  IMRT external beam pelvic radiation therapy as appropriate for stage
  Intracavitary brachytherapy (6 HDR treatments)
  Weekly cisplatin (40 mg/m^2)
Period: Overall Study
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Started | 44 | 25
Completed | 41 | 20
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Ineligible | 1 | 0
Not completed — Poor performance status | 0 | 1
Not completed — Non-compliant | 0 | 2
Not completed — Did not sign consent form | 0 | 1
Not completed — Did not receive chemo per protocol | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group 1 (IMRT, Brachytherapy, Cisplatin): Pelvic Lymph Nodes Only Positive on FDG PET.
  IMRT External Beam radiation to the para-aortic region (45 Gy)
  Pelvis intracavitary brachytherapy (6 HDR treatments)
  Weekly cisplatin 40 mg/m^2
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin) | Total
Number analyzed (Participants) | 41 | 20 | 61
Age, Continuous [Median (Full Range); unit: years] | 45 [26 to 77] | 52 [39 to 62] | 45 [26 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 20 | 61
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Tolerance of IMRT Extended-field External Radiotherapy to Pelvis and Para-aortic Region, Combined With Intracavitary Irradiation, and Cisplatin Chemotherapy as Measured the Number of Participants With by Grade 4 or Higher Toxicity
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for all toxicity reporting.
Time Frame: 1 year post start of radiation therapy
Measure: Number; unit: participants
Groups:
- Treatment Group 1 (IMRT, Brachytherapy, Cisplatin): Pelvic Lymph Nodes Only Positive on FDG PET.
  IMRT External Beam radiation to the para-aortic region (45 Gy)
  Pelvis intracavitary brachytherapy (6 HDR treatments)
  Weekly cisplatin (40 mg/m^2)
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Number analyzed (Participants) | 41 | 20
participants
  Neutropenia | 3 | 1
  Anorexia | 1 | 1
  Diarrhea | 1 | 1
  Hypomagnesemia | 1 | 0
  Leukopenia | 2 | 3
  Lymphopenia | 1 | 3
  Dyspnea | 0 | 1
  Fatigue | 0 | 1
  Hemoglobin | 0 | 2
  Hematocrit | 0 | 1
  Hyperkalemia | 0 | 1
  Hypoglycemia | 0 | 1
  Hyponatremia | 0 | 1
  Infection without neutropenia | 0 | 1
  Platelets | 0 | 1
  Renal failure | 0 | 1

2. Primary Outcome: Number of Participants With Acute Toxicity of IMRT Extended-field External Radiotherapy to Pelvis and Para-aortic Region, Combined With Intracavitary Irradiation, and Cisplatin Chemotherapy (Grade 3 or Higher)
Time Frame: 30 days after completion of radiation therapy
Measure: Number; unit: participants
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Number analyzed (Participants) | 41 | 20
participants
  Absolute neutrophil count | 6 | 4
  Anorexia | 1 | 1
  Anxiety | 1 | 0
  Diarrhea | 5 | 5
  Dyspnea | 1 | 1
  Dysuria | 1 | 0
  Fatigue | 9 | 4
  Granulocytes/bands | 1 | 2
  Hemoglobin | 2 | 6
  Hematocrit | 1 | 4
  Vaginal bleeding | 1 | 0
  Hyperglycemia | 1 | 1
  Hypermagnesemia | 1 | 0
  Hypertension | 2 | 0
  Hypocalcemia | 3 | 0
  Hypokalemia | 5 | 0
  Hyponatremia | 3 | 4
  Hypomagnesemia | 1 | 5
  Infection with neutropenia | 1 | 2
  Infection (Urinalysis) | 1 | 3
  Leukopenia | 10 | 10
  Lymphopenia | 35 | 25
  Nausea | 4 | 1
  Abdominal pain | 3 | 1
  Pelvic pain | 2 | 2
  Pain - not otherwise specified (NOS) | 4 | 0
  packed red blood cell (PRBC) Transfusion | 5 | 11
  Platelets | 2 | 2
  Proteinuria | 1 | 0
  Skin | 1 | 2
  Vomiting | 2 | 1
  Weight loss | 2 | 2
  Albumin | 0 | 1
  Atrial fibrillation | 0 | 1
  Confusion | 0 | 1
  Creatinine | 0 | 1
  Vaginal mucosa erythematous | 0 | 1
  Edema | 0 | 1
  erythrocyte sedimentation rate (ESR) | 0 | 1
  Hyperkalemia | 0 | 1
  Hypoglycemia | 0 | 2
  international normalized ratio (INR) | 0 | 1
  Leucocyte esterase | 0 | 1
  Prothrombin time (PT) | 0 | 1
  partial thromboplastin time (PTT) | 0 | 4
  Renal failure | 0 | 1
  aspartate aminotransferase (ALT) | 0 | 1
  Yeast infection | 0 | 1

3. Primary Outcome: Efficacy of IMRT Extended-field Radiation Combined With Intracavitary Irradiation, and Cisplatin Chemotherapy as Measured by PET Scan Disease Status
Time Frame: 1st PET scan after completion of treatment (approximately month 6)
Measure: Number; unit: participants
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Number analyzed (Participants) | 41 | 20
participants
  Positive PET scan | 6 | 9
  Negative PET scan | 27 | 7
  Equivocal PET scan | 6 | 4
  PET scan not performed | 2 | 0

4. Secondary Outcome: Efficacy of IMRT to the Para-aortic Lymph Nodes, IMRT External Beam Radiotherapy to the Pelvis, Intracavitary Irradiation, and Cisplatin Chemotherapy as Measured by the Frequency of Distant Metastasis
Time Frame: 5 years after completion of radiation therapy
Population: The data was not collected for this secondary outcome. Due to the the early termination of this study, only data for the primary outcomes were collected and analyzed.
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Serious adverse events are events that had serious adverse event reports filed with the institutional review board.
Arm/Group | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin)
Serious Adverse Events (participants affected / at risk) | 10/41 | 4/20
Other Adverse Events (participants affected / at risk) | 41/41 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) (N=41) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin) (N=20)
Hypertension (Vascular disorders) | 1 | 0
Fever (General disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 6 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Infection without neutropenia (Infections and infestations) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Investigations) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (ANC) (Investigations) | 1 | 0
Lymphopenia (Investigations) | 1 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 | 0
Skin pain (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Rigors/chills (General disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Polymicrobial sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (IMRT, Brachytherapy, Cisplatin) (N=41) | Treatment Group 2 (IMRT, Brachytherapy, Cisplatin) (N=20)
Abdominal pain (Gastrointestinal disorders) | 9 | 4
Absolute neutrophil count (ANC) (Investigations) | 10 | 11
Albumin (Metabolism and nutrition disorders) | 3 | 3
Alkaline phosphatase (Investigations) | 4 | 6
Anorexia (Metabolism and nutrition disorders) | 16 | 16
Anxiety (Psychiatric disorders) | 4 | 5
Atrial Fibrillation (Cardiac disorders) | 1 | 1
BUN (Investigations) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bilirubin (Investigations) | 6 | 6
CO2 (elevated) (Investigations) | 6 | 3
Cardiac dysrhythmias (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 1
Chills (General disorders) | 2 | 1
Chloride (Investigations) | 4 | 1
Confusion (Psychiatric disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine (Investigations) | 7 | 9
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 3
Dermatologic (vaginal mucosa erythematous) (Skin and subcutaneous tissue disorders) | 9 | 10
Diarrhea (Gastrointestinal disorders) | 33 | 20
Dizziness (Nervous system disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dysuria (Renal and urinary disorders) | 9 | 6
Edema (General disorders) | 2 | 5
Fatigue (General disorders) | 28 | 19
Fever (General disorders) | 3 | 2
Granulocytes/Bands (Investigations) | 4 | 5
Hematologic - other (RBCs) (Blood and lymphatic system disorders) | 1 | 1
Hematologic - other (hematocrit) (Blood and lymphatic system disorders) | 5 | 7
Hematuria (Renal and urinary disorders) | 8 | 7
Hemoglobin (Blood and lymphatic system disorders) | 33 | 20
Hemorrhage (rectal bleeding) (Gastrointestinal disorders) | 1 | 1
Hemorrhage (vaginal bleeding) (Reproductive system and breast disorders) | 3 | 2
Hemorrhagic cystitis (Renal and urinary disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyperproteinemia (Metabolism and nutrition disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 3
Hypobilirubinemia (Investigations) | 2 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 12
Hypokalemia (Metabolism and nutrition disorders) | 18 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 10
Hyponatremia (Metabolism and nutrition disorders) | 11 | 12
Hypotension (Vascular disorders) | 6 | 1
Infection (Respiratory) (Infections and infestations) | 1 | 0
Infection (urinalysis) (Infections and infestations) | 8 | 6
Infection with neutropenia (Infections and infestations) | 1 | 2
LDH (Investigations) | 2 | 0
Leucocyte esterase (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Investigations) | 27 | 19
Lymphopenia (Investigations) | 36 | 20
Nausea (Gastrointestinal disorders) | 31 | 20
Neuro-mood (Psychiatric disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 2 | 1
PRBC Transfusion (Blood and lymphatic system disorders) | 5 | 11
PT (Investigations) | 3 | 6
PTT (Investigations) | 5 | 4
Pain NOS (General disorders) | 7 | 3
Pelvic pain (Reproductive system and breast disorders) | 8 | 6
Plasma Protein (Investigations) | 1 | 0
Platelets (Investigations) | 17 | 15
Proteinuria (Renal and urinary disorders) | 6 | 6
Rectal pain (Gastrointestinal disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
SGOT (Investigations) | 5 | 3
SGPT (Investigations) | 3 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 0
Skin (Skin and subcutaneous tissue disorders) | 22 | 16
Sun intolerance (Skin and subcutaneous tissue disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 11 | 10
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 19 | 12
Weight loss (Investigations) | 21 | 10
Dermatologic (local) (Skin and subcutaneous tissue disorders) | 0 | 1
Dyphagia/esophagitis (Gastrointestinal disorders) | 0 | 1
ESR (Blood and lymphatic system disorders) | 0 | 1
Gastrointestinal (heartburn) (Gastrointestinal disorders) | 0 | 1
INR (Investigations) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Memory loss (Nervous system disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Yeast infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes